CLINICAL TRIAL: NCT02276872
Title: A Multicenter, Open-Label, 24-Week, Uncontrolled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral Treprostinil Extended Release Tablets Following Transition From Remodulin or Inhaled Prostacyclin Therapy or as Add-on to Current PAH Therapy in De Novo Prostacyclin Pediatric Subjects Aged 7 to 17 Years With Pulmonary Arterial Hypertension
Brief Title: Safety, Tolerability, and Pharmacokinetics of Oral Treprostinil in Pediatric PAH Patients Aged 7 to 17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-206
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: PAH
Keywords: pediatric; treprostinil; transition; Remodulin
MeSH Terms: interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Transitioning from Parental) (Experimental): Transitioned from IV or SC Remodulin to oral treprostinil
  Interventions: Drug: oral treprostinil
- Cohort 2 (Transitioning from Inhaled) (Experimental): Transitioned from inhaled prostacyclin to oral treprostinil
  Interventions: Drug: oral treprostinil
- Cohort 3 (Add-on to Current PAH Therapy) (Experimental): Treated with oral treprostinil as a de novo add-on to current PAH therapy
  Interventions: Drug: oral treprostinil

INTERVENTIONS:
Drug: oral treprostinil
  Other Names: Orenitram

SUMMARY:
This was a multi-center, open-label, safety, tolerability and pharmacokinetic study of oral treprostinil in pediatric subjects with stable PAH aged 7 to 17 years who were (1) transitioning from parenteral Remodulin therapy; (2) transitioning from inhaled prostacyclin therapy; or (3) not currently receiving prostacyclin therapy.

DETAILED DESCRIPTION:
Study TDE-PH-206 was a multicenter, open-label study designed to investigate the safety, tolerability, and PK of oral treprostinil administered 3 times daily (TID) or 4 times daily (QID), at the discretion of the Investigator, with food in pediatric PAH subjects aged 7 to 17 years of age (1) transitioning from continuous IV/SC Remodulin, (2) transitioning from inhaled prostacyclin, or (3) as add-on to current PAH therapies in de novo prostacyclin subjects. Eligible subjects were assigned to a cohort based upon their background therapy. All subjects received oral treprostinil provided as 0.125, 0.25, 1, or 2.5 mg extended-release tablets. Subjects in Cohort 1 began the transition from IV/SC Remodulin in the hospital with a goal of complete transition to oral treprostinil within 5 days. The initial dose of oral treprostinil for Cohort 1 was calculated from the subject's dose of IV/SC Remodulin and weight. Subjects in Cohorts 2 and 3 were initiated on 0.125 mg TID or QID oral treprostinil with dose escalations possible every 24 hours in increments of 0.125 mg TID or QID at the discretion of the Investigator during the first 4 weeks, and in increments of either 0.125 mg or 0.25 mg every 24 hours thereafter. Cross titration occurred for Cohorts 1 and 2 such that doses of IV/SC Remodulin or inhaled prostacyclin were decreased as subjects were fully transitioned to oral treprostinil.

ELIGIBILITY:
Inclusion Criteria:

1. Legal guardian informed consent and subject assent, if appropriate, to participate in the study was voluntarily given.
2. The subject was between 7 and 17 years of age, inclusive, on the date informed consent was signed.
3. Cohort 3: The subject weighed a minimum of 22 kg at Screening.
4. The subject had a current diagnosis of PAH (WHO Group I) associated with:

   1. IPAH or HPAH
   2. Persistent PAH for at least 1 year following surgical repair of a congenital systemic-to-pulmonary cardiac shunt, congenital heart disease, or other congenital heart lesions with no clinically significant residual defects and condition was stabilized hemodynamically
   3. PAH in subjects with unrepaired restricted atrial septal defect, ventricular septal defect, or patent ductus arteriosus; subject had a resting post-ductal oxygen saturation (off oxygen) of greater than 88%.
5. The subject had a current diagnosis of PAH confirmed by RHC prior to the Screening Visit with the following parameters:

   1. PAPm of ≥25 mmHg
   2. Pulmonary vascular resistance index (PVRi) of >3 Wood Units*m2
   3. Left ventricular end-diastolic pressure (LVEDP) or pulmonary capillary wedge pressure (PCWP) of ≤15 mmHg.
6. Cohort 1: The subject had received IV/SC Remodulin for at least 90 days without dose change for at least 30 days prior to Baseline. The IV/SC Remodulin dose was between 25 to 75 ng/kg/min, inclusive, for the first 5 subjects in the cohort. Following safety review, the dose range was expanded to 25 to 125 ng/kg/min, inclusive, for the remaining subjects. Subjects must have received stable doses of all other PAH medications for at least 14 days prior to the baseline assessments; exception for diuretics and anticoagulants.
7. Cohort 2: The subject must have received inhaled prostacyclin for at least 90 days and had been at the current stable dose without changes for at least 30 days prior to Baseline. Subjects must have received stable doses of all other PAH medications for at least 14 days prior to the baseline assessments; exception for diuretics and anticoagulants.
8. All Cohorts: All subjects were optimally treated (as determined by the Investigator) with background PAH therapies (eg, phosphodiesterase type 5 inhibitor [PDE5-I], endothelin receptor antagonist [ERA], soluble guanylate cyclase [sGC]) for at least 90 days and had been on a stable dose without changes (except documented weight based adjustments) for at least 30 days prior to the first dose of oral treprostinil. Subjects must have received stable doses of all other PAH medications for at least 14 days prior to the first dose of oral treprostinil; exception for diuretics and anticoagulants.
9. The subject was willing and able to swallow intact tablets whole without chewing, breaking, or splitting.
10. The subject was willing and able to comply with the dietary requirements associated with the oral treprostinil dosing regimen.
11. The subject was on stable doses of other medical therapy for 14 days prior to the Baseline Visit with no dose adjustments, additions, or discontinuations. Dose changes of diuretics were allowed if within the usual dose adjustments prescribed for the subject. Anticoagulants could have been adjusted, but not discontinued or added, within 14 days of Baseline. Temporary discontinuation of anticoagulants when related to study-related procedures was allowed.
12. Females of childbearing potential include any female who had experienced menarche. Females of childbearing potential must have practiced true abstinence from intercourse, had an intrauterine device, or used 2 different forms of highly effective contraception for the duration of the study and for at least 30 days after discontinuing oral treprostinil. Medically acceptable forms of effective contraception included approved hormonal contraceptives (such as birth control pills) or barrier methods (such as a condom or diaphragm) used with a spermicide. For females of childbearing potential, a negative urine pregnancy test was required at Baseline prior to oral treprostinil administration. Males participating in the study must have used a condom during intercourse for the duration of the study and for at least 48 hours after discontinuing oral treprostinil.
13. Subjects with a history of metallic implants, prior neurosurgical clip placement, or other potential contraindications to cMRI were individually evaluated per site standard operating procedures for MRI performance.
14. In the opinion of the Principal Investigator, the subject and/or legal guardian was able to communicate effectively with study personnel, and was considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. The subject had a diagnosis of large unrestrictive ventricular septal defect or patent ductus arteriosus, Eisenmenger syndrome, congenital diaphragmatic hernia, or a chronic lung disease, such as bronchopulmonary dysplasia or interstitial lung disease.
2. The subject had a current disease severity of Panama FC IIIb or IV.
3. The subject had previously been exposed to oral treprostinil.
4. Cohort 1: The subject had previous intolerance to treprostinil or epoprostenol due to systemic adverse effects that resulted in discontinuation of therapy. This did not include site pain reactions or central venous catheter-related blood stream infections.
5. Cohort 1 and 2: The subject was receiving IV/SC Remodulin or Tyvaso® (as the inhaled prostacyclin) for any other disease or condition other than the treatment of PAH in accordance with the IV/SC Remodulin or Tyvaso package inserts (ie, eligible subjects must have had a WHO Group I PAH classification as defined in inclusion criterion #4).
6. Cohort 3: The subject had been previously exposed to a prostacyclin within 30 days of Screening, with the exception of vasoreactivity testing.
7. The subject was pregnant or lactating.
8. The subject had a current diagnosis of uncontrolled sleep apnea as defined by their physician.
9. The subject had severe renal insufficiency as defined by an estimated creatinine clearance <30 mL/min (Schwartz Formula) or the requirement for dialysis at Screening.
10. The subject had moderate to severe hepatic dysfunction as defined by elevated liver function tests (aspartate aminotransferase or alanine aminotransferase) ≥3 times the upper limit of normal at Screening, or Child Pugh class B or C hepatic disease.
11. The subject had clinically significant anemia as defined by a hemoglobin and/or hematocrit level <75% of the lower limit of normal ranges according to age and gender.
12. The subject had Down Syndrome.
13. The subject had uncontrolled systemic hypertension as evidenced by a systolic or diastolic blood pressure greater than the 95th percentile for age, height, and gender at Screening or Baseline.
14. The subject and/or legal guardian had an unstable psychiatric condition or was mentally incapable of understanding the objectives, nature, or consequences of the study, or had any condition in which the Investigator's opinion would constitute an unacceptable risk to the subject's safety.
15. The subject had an active infection or any other cardiovascular, liver, renal, hematologic, gastrointestinal, immunologic, endocrine, metabolic, or central nervous system disease or condition that, in the opinion of the Investigator, might have adversely affected the safety of the subject or interfered with the interpretation of study assessments.
16. Subject was actively listed for transplantation.
17. The subject was receiving an investigational drug, had an investigational device in place, or had participated in an investigational drug or device study within 30 days prior to Baseline. Participation in an observational study did not disqualify a potential subject from study participation.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dunbar Ivy, MD, Principal Investigator — Denver Children's Hospital
Locations (9):
- United States (9):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Ivy DD, Feinstein JA, Yung D, Mullen MP, Kirkpatrick EC, Hirsch R, Austin ED, Fineman J, Truong U, Solum D, Deng CQ, Hopper RK. Oral treprostinil in transition or as add-on therapy in pediatric pulmonary arterial hypertension. Pulm Circ. 2019 Jul-Sep;9(3):2045894019856471. doi: 10.1177/2045894019856471. PMID 31215336
- [Background] Hopper RK, Ivy DD, Yung D, Mullen MP, Hanna BD, Kirkpatrick E, Hirsch R, Austin ED, Fineman J, Solum D, Deng CQ, Feinstein JA. Pharmacokinetics of Oral Treprostinil in Children With Pulmonary Arterial Hypertension. J Cardiovasc Pharmacol. 2020 Jul;76(1):94-100. doi: 10.1097/FJC.0000000000000842. PMID 32398473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Started | 10 | 10 | 12
Completed | 9 | 10 | 12
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy) | Total
Number analyzed (Participants) | 10 | 10 | 12 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 12 | 32
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10.0 [7 to 17] | 13.5 [8 to 17] | 13.5 [8 to 17] | 12 [7 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 7 | 23
  Male | 1 | 3 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 7
  Not Hispanic or Latino | 6 | 8 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 9 | 10 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Transition From IV/SC Remodulin to Oral Treprostinil (Cohort 1), From Inhaled Prostacyclin to Oral Treprostinil (Cohort 2), or as an add-on to Current PAH Therapy in de Novo Prostacyclin Subjects (Cohort 3).
Description: A successful transition was defined as a subject from Cohort 1 or Cohort 2 who was receiving oral treprostinil and no longer receiving IV/SC Remodulin or inhaled prostacyclin, respectively, at Week 4 and clinically maintained on oral treprostinil treatment through Week 24. A successful initiation of oral treprostinil for Cohort 3 was defined as a subject who was clinically maintained on oral treprostinil through Week 24.
Time Frame: Up to 24 weeks
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 10 | 10 | 12
participants
  Successfully transitioned/initiated within 4 weeks | 10 | 10 | 12
  Successfully maintained through 24 weeks | 9 | 10 | 12

2. Secondary Outcome: Cardiopulmonary Exercise Testing - Change From Baseline in Peak Oxygen Uptake (VO2) at Week 24
Description: Cardiopulmonary Exercise Testing (CPET) was performed with progressive cycle ergometry and ventilatory expired gas analysis obtained using a metabolic cart at Baseline and Week 24/Premature Termination. CPET consisted of measuring oxygen uptake (VO2), carbon dioxide output (VCO2), minute ventilation (VE), and other variables in addition to a 12-lead ECG, blood pressure (BP) monitoring, and pulse oximetry.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Testing at Week 24
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 5 | 9 | 12
mL/kg/min | -3.26 (7.34) | 2.18 (8.01) | 2.00 (3.47)

3. Secondary Outcome: Cardiopulmonary Exercise Testing - Change From Baseline in Minute Ventilation (VE)/Carbon Dioxide Output (VCO2) Slope at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Testing at Week 24
Measure: Mean (Standard Deviation); unit: VE/VCO2 Slope
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 5 | 9 | 12
VE/VCO2 Slope | -1.066 (3.169) | 2.170 (5.111) | 1.531 (3.821)

4. Secondary Outcome: Cardiopulmonary Exercise Testing - Change From Baseline in Peak Watts at Week 24
Description: as for outcome 2
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Testing at Week 24
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 6 | 9 | 11
Watts | 4.8 (10.3) | -2.8 (11.9) | 6.5 (12.9)

5. Secondary Outcome: Change in Symptoms of PAH From Baseline to Week 24
Description: PAH symptoms (fatigue, dyspnea, edema, dizziness, syncope, chest pain, orthopnea) were assessed at the Baseline Visit prior to the initiation of oral treprostinil dosing and at Week 24. Scores range from 0 (for the best condition) to 3 (for the worst condition).
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
Participants
  Chest Pain - Improved - Week 24 | 0 | 0 | 2
  Chest Pain - No Change - Week 24 | 8 | 9 | 8
  Chest Pain - Deteriorated - Week 24 | 1 | 1 | 2
  Dizziness - Improved - Week 24 | 0 | 0 | 4
  Dizziness - No Change - Week 24 | 9 | 8 | 8
  Dizziness - Deteriorated - Week 24 | 0 | 2 | 0
  Dyspnea - Improved - Week 24 | 3 | 0 | 5
  Dyspnea - No Change - Week 24 | 4 | 8 | 6
  Dyspnea - Deteriorated - Week 24 | 2 | 2 | 1
  Edema - Improved - Week 24 | 0 | 0 | 1
  Edema - No Change - Week 24 | 8 | 10 | 10
  Edema - Deteriorated - Week 24 | 1 | 0 | 1
  Fatigue - Improved - Week 24 | 0 | 3 | 2
  Fatigue - No Change - Week 24 | 5 | 6 | 9
  Fatigue - Deteriorated - Week 24 | 4 | 1 | 1
  Orthopnea - Improved - Week 24 | 0 | 0 | 3
  Orthopnea - No Change - Week 24 | 9 | 10 | 9
  Orthopnea - Deteriorated - Week 24 | 0 | 0 | 0

6. Secondary Outcome: Change in Panama Functional Class From Baseline to Week 24
Description: Change from Baseline in subject clinical status was recorded according to the Panama Functional Class.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
Participants
  Improved - Week 24 | 0 | 2 | 3
  No Change - Week 24 | 9 | 7 | 9
  Deteriorated - Week 24 | 0 | 1 | 0

7. Secondary Outcome: Change in WHO Functional Class From Baseline to Week 24
Description: Change from Baseline in subject clinical status was recorded according to the WHO Functional Class.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
Participants
  Improved - Week 24 | 0 | 1 | 3
  No Change - Week 24 | 9 | 8 | 9
  Deteriorated - Week 24 | 0 | 1 | 0

8. Secondary Outcome: Change in 6-Minute Walk Distance (6MWD) From Baseline to Week 24
Description: The intent of the 6MWT was to evaluate exercise capacity associated with carrying out activities of daily living. Total distance covered in a total of 6 minutes was measured. Oxygen saturation and heart rate (HR) were measured at rest prior to the 6MWT and monitored continuously during the walk. Recovery monitoring (HR and oxygen saturation) was performed and documented at Minute 0 (immediately upon stopping the 6MWT), Minute 1, Minute 2, and Minute 3 post walk.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
meters | 2.7 (94.2) | 22.1 (86.5) | 12.8 (49.6)

9. Secondary Outcome: Change in Borg Dyspnea Score From Baseline to Week 24
Description: The Borg dyspnea score was assessed prior to and following the completion of the 6MWT at Week 24. The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6MWT. Scores range from 0 (for the best condition) to 10 (for the worst condition).
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort 1 (Transitioning From Parental): Transitioned from IV or SC Remodulin to oral treprostinil
  oral treprostinil
- Cohort 2 (Transitioning From Inhaled): Transitioned from inhaled prostacyclin to oral treprostinil
  oral treprostinil
- Cohort 3 (Add-on to Current PAH Therapy): Treated with oral treprostinil as a de novo add-on to current PAH therapy
  oral treprostinil
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
score on a scale | -1.56 (3.51) | 0.05 (1.50) | -0.83 (1.59)

10. Secondary Outcome: Change in Quality of Life Assessed Via the Pediatric Quality of Life Inventory (PedsQL) Questionnaire From Baseline to Week 24
Description: Four subscales [items]: (Physical [8], Emotional [5], Social [5], School Functioning [5]). Subjects and subjects' parent(s) completed PedsQL at Week 24. Response to each item on the subscales were graded 0-4 (0=never a problem, 1=almost never a problem, 2=sometimes a problem, 3=often a problem, 4=almost always a problem). Response to each item was transformed from the 0-4 scale to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Using transformed values, mean was computed as sum of the items in each subscale over number of items answered in the same subscale. Two summary scores (Psychosocial Health Summary Score and Total Scale Score) were calculated with a range of 0-100 (higher values indicating better outcome). Psychosocial Health Summary Score was mean computed as sum of the items over the number of items answered in the Emotional, Social, and School Functioning Scales. Total Score was calculated as sum of all items over number of items answered on all the scales.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
score on a scale
  Physical Functioning - Child - Week 24 | 5.57 (22.14) | -2.82 (11.09) | 5.48 (13.40)
  Emotional Functioning - Child - Week 24 | 8.33 (11.46) | 3.00 (13.98) | 2.92 (13.05)
  Social Functioning - Child - Week 24 | 9.44 (16.85) | 0.00 (15.09) | 1.25 (11.31)
  School Functioning - Child - Week 24 | 3.89 (23.29) | -6.50 (11.56) | 7.92 (21.37)
  Psychosocial Health - Child - Week 24 | 7.23 (13.52) | -1.17 (11.11) | 4.04 (11.85)
  Total Scale Score - Child - Week 24 | 6.64 (15.08) | -1.76 (8.54) | 4.53 (11.46)
  Physical Functioning - Parent - Week 24 | 1.72 (12.31) | -2.81 (14.98) | 1.29 (14.67)
  Emotional Functioning - Parent - Week 24 | -2.22 (15.63) | 2.50 (10.07) | 5.00 (18.95)
  Social Functioning - Parent - Week 24 | -1.11 (14.53) | -5.50 (18.92) | 11.67 (16.28)
  School Functioning - Parent - Week 24 | 9.44 (16.85) | -5.50 (11.65) | 5.00 (13.14)
  Psychosocial Health - Parent - Week 24 | 2.04 (13.80) | -2.81 (11.48) | 7.22 (13.21)
  Total Scale Score - Parent - Week 24 | 1.93 (11.79) | -2.84 (12.29) | 5.17 (12.78)

11. Secondary Outcome: Change in Plasma N-terminal Pro-B-type Natriuretic Peptide (NT-Pro BNP) From Baseline to Week 24
Description: Plasma NT-proBNP concentration is a useful biomarker for PAH as it is associated with changes in right heart morphology and function.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects that Completed Study Week 24
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 9 | 10 | 12
pg/mL | 87.156 (281.664) | 81.930 (245.534) | 160.617 (549.953)

12. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Week 24
Description: Cardiac MRI imaging was performed in all subjects aged 10 years and older at Baseline and Week 24/Premature Termination; imaging was optionally performed in subjects under the age of 10 years. The subject's BP was taken immediately prior to the cMRI assessment in the supine position to measure vascular parameters.
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
percentage of LVEF | -1.0 (1.4) | 2.4 (6.0) | -2.4 (3.1)

13. Secondary Outcome: Change From Baseline in Left Ventricular (LV) Stroke Volume Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: mL/beat/m2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
mL/beat/m2 | -4.003 (2.688) | 6.336 (8.448) | 1.113 (5.539)

14. Secondary Outcome: Change From Baseline in Right Ventricular (RV) Cardiac Output Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: L/min/m2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
L/min/m2 | 0.303 (0.209) | 0.767 (1.010) | 0.121 (1.047)

15. Secondary Outcome: Change From Baseline in Right Ventricular End-diastolic Volume (RVEDV) Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: mL/m^2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
mL/m^2 | -8.190 (12.887) | 12.131 (14.382) | 10.601 (26.115)

16. Secondary Outcome: Change From Baseline in Right Ventricular Ejection Fraction (RVEF) at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: percentage of RVEF
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
percentage of RVEF | 4.0 (7.6) | 0.4 (7.1) | -0.7 (2.7)

17. Secondary Outcome: Change From Baseline in Right Ventricular End-systolic Volume (RVESV) Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: mL/m2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
mL/m2 | -7.975 (12.614) | 5.884 (12.965) | 5.722 (13.807)

18. Secondary Outcome: Change From Baseline in Right Ventricular (RV) Mass Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: g/m2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
g/m2 | 2.375 (6.226) | 3.041 (7.890) | 0.614 (3.450)

19. Secondary Outcome: Change From Baseline in Right Ventricular (RV) Stroke Volume Index at Week 24
Description: as for outcome 12
Time Frame: Baseline and Week 24
Population: Safety Population - Number of Subjects with both Baseline and Week 24 Measurements
Measure: Mean (Standard Error); unit: mL/beat//m2
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
Number analyzed (Participants) | 4 | 9 | 9
mL/beat//m2 | -0.215 (1.557) | 6.193 (8.015) | 1.458 (6.719)

20. Secondary Outcome: Maximum Observed Drug Concentration in Plasma (Cmax)
Description: Cohort 1 had three blood samples obtained at 'Time 0' and at 4 and 8 hours at the Baseline visit. All cohorts had five blood samples obtained from at 'Time 0' and at 2, 4, 6, and 8 hours at the Week 24 visit. Plasma samples were analyzed for treprostinil using a validated bioanalytical plasma assay. Individual and mean treprostinil plasma concentration data and treprostinil pharmacokinetic parameters, such as peak observed plasma concentration (Cmax), time to peak plasma concentration (Tmax), area under the plasma concentration-time curve (AUC0-inf), were determined as able. For the purposes of PK analysis, data for Cohorts 1, 2, and 3 following oral treprostinil administration were combined and compared to parenteral infusion (Cohort 1 Baseline data; Remodulin IV/SC).
Time Frame: Baseline (Cohort 1 only; 0, 4, 8 hours while receiving IV/SC Remodulin) and Week 24 (all cohorts; 0, 2, 4, 6, 8 hours post-dose oral treprostinil)
Population: PK Population. To provide a larger sample size for PK analysis, data for Cohorts 1, 2, and 3 following oral treprostinil administration were combined and compared to parenteral infusion (Cohort 1 Baseline data; Remodulin IV/SC).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort 1 (Transitioning From Parenteral): Transitioned from IV or SC Remodulin to oral treprostinil
- Cohorts Combined After Oral Treprostinil Administration: Combined PK data for Cohorts 1, 2, and 3 combined after oral treprostinil administration
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
ng/mL | 5.14 (39.4) | 4.91 (50.5)

21. Secondary Outcome: Last Observed Drug Concentration in Plasma (Clast)
Description: Cohort 1 had three blood samples obtained at 'Time 0' and at 4 and 8 hours at the Baseline visit. All cohorts had five blood samples obtained from at 'Time 0' and at 2, 4, 6, and 8 hours at the Week 24 visit. Plasma samples were analyzed for treprostinil using a validated bioanalytical plasma assay. Individual and mean treprostinil plasma concentration data and treprostinil pharmacokinetic parameters, such as peak observed plasma concentration (Cmax), time to peak plasma concentration (Tmax), area under the plasma concentration-time curve (AUC0-inf), were determined as able.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
ng/mL | 4.66 (38.6) | 0.985 (104)

22. Secondary Outcome: Average Drug Concentration in Plasma (Cavg)
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
ng/mL | 4.28 (37.7) | 2.80 (54.5)

23. Secondary Outcome: Observed Minimum Drug Concentration in Plasma (Cmin)
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
ng/mL | 3.45 (47.9) | 0.799 (88.5)

24. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to Tau Hours Post-dose (AUCtau)
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
h*ng/mL | 34.3 (37.7) | 22.2 (53.8)

25. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to 8 Hours Post-dose (AUC0-8)
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 (Transitioning From Parenteral) | Cohorts Combined After Oral Treprostinil Administration
Number analyzed (Participants) | 10 | 32
h*ng/mL | 34.3 (37.7) | 22.4 (54.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time that each subject and/or caregiver signed the ICF until the time screen failure was documented, or until the subject was either discontinued from the study or all Week 24 study assessments were completed.
Arm/Group | Cohort 1 (Transitioning From Parental) | Cohort 2 (Transitioning From Inhaled) | Cohort 3 (Add-on to Current PAH Therapy)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/10 | 0/10 | 4/12
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Transitioning From Parental) (N=10) | Cohort 2 (Transitioning From Inhaled) (N=10) | Cohort 3 (Add-on to Current PAH Therapy) (N=12)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Transitioning From Parental) (N=10) | Cohort 2 (Transitioning From Inhaled) (N=10) | Cohort 3 (Add-on to Current PAH Therapy) (N=12)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Excessive eye blinking (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Perioribital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 9 (10)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (6) | 9 (9)
Vomiting (Gastrointestinal disorders) | 9 (9) | 5 (6) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 4 (4) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 5 (6)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (5) | 2 (2)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 2 (2) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 8 (9) | 12 (12)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 4 (4)
Syncope (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Periodic limb movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intentional self injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 6 (6) | 4 (4) | 8 (8)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02276872/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02276872/SAP_000.pdf